CLINICAL TRIAL: NCT05419739
Title: Prognostic Value of Pediatric GCS-Pupil Score in Pediatric Patients With Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, AKİF BULUT, Principal Investigator, Uludag University
Other Study IDs: 2011-KAEK-25 2022/04-08
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Brain Injuries, Traumatic
Keywords: Brain traumatic; GCS-Pupil score; Pediatric
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Glasgow Coma Scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Children under 18 years of age with traumatic brain injury
  Interventions: Other: Glasgow coma scale

INTERVENTIONS:
Other: Glasgow coma scale — This scale, which consists of three parameters, includes the best eye response (1-4 points), the best verbal response (1-5 points), and the best motor response (1-6 points). Total score; It is calculated as Eye Response + Verbal Response + Motor Response and takes a value between 3-15 points. The severity of head trauma is evaluated in three categories: mild (GCS 13-15 points), moderate (GCS 9-12 points), and severe (GCS ≤ 8 points).
  Other Names: Pediatric Cerebral Performance Category Scoring System

SUMMARY:
There are studies reporting that the survival rate in pediatric patients with abnormal pupillary response is 23% and that pupillary response is effective on mortality and patient outcomes. Studies in the literature examining the effect of pupillary response on mortality and outcome in pediatric patients with traumatic brain injury reported that bilaterally dilated pupils were associated with a higher mortality rate.

Considering the literature results, we believe that obtaining the GCS-Pupil score by combining GCS and pupillary reaction in pediatric patients with traumatic brain injury will be effective in predicting patient outcomes.

DETAILED DESCRIPTION:
Obtaining a GCS-Pupil score using the total GCS score: 0 points are given for pupillary reaction if both pupils react to light, 1 point if one pupil does not react to light, and 2 points if both pupils do not react to light. Total GCS-P score is calculated by the formula of Eye Response + Verbal Response + Motor Response - Pupil Reaction and scores between 1-15.

In the study, the worst GCS and current pupillary light reaction score in the first 24 hours will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Be under the age of 18,
* Not having mental and motor developmental retardation,
* Having had a traumatic brain injury,
* Alive at admission and followed up for at least 24 hours

Exclusion Criteria:

* Eye trauma or severe facial trauma that will affect the assessment,
* Those under deep sedation,
* Those who have been administered drugs (Atropine and mydriatic) that will affect the pupillary response.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients younger than 18 years with traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Death rate | one year
  Death

SECONDARY OUTCOMES:
Adverse functional outcomes | one year
  severely crippled or vegetative condition

CONTACTS AND LOCATIONS:
Overall Officials: AKİF BULUT, MSc, Principal Investigator — Uludag University
Locations (1):
- Bursa Provincial Health Directorate University of Health Sciences Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers.